CLINICAL TRIAL: NCT04160390
Title: Blood Samples to Identify Biomarkers for Post-Transplant Cyclophosphamide
Brief Title: Blood Samples to Identify Biomarkers in Patients Treated With Cyclophosphamide After Donor Stem Cell Transplant
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18358; NCI-2019-07376 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18358 (Other: City of Hope Medical Center); U01CA239373 (NIH)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplant Recipient; Donor; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm I (biospecimen collection): Patients undergo collection of blood prior to transplant, on day 0, days 3-7, day 14, and day 21. Patients also undergo collection of saliva prior to transplant and collection of stool prior to and post-transplant. Donors undergo collection of blood and saliva within 8 weeks prior to donation.
  Interventions: Other: Biospecimen Collection-Blood; Other: Biospecimen Collection-Stool

INTERVENTIONS:
Other: Biospecimen Collection-Blood — Undergo collection of blood
Other: Biospecimen Collection-Stool — Undergo collection of stool

SUMMARY:
This trial uses blood samples to understand how patients' bodies process and respond to a drug called cyclophosphamide given after a donor stem cell transplant. Identifying biomarkers (molecules that can indicate normal or abnormal processes) may help researchers develop a blood test that can be used to predict how well patients will process and respond to cyclophosphamide.

DETAILED DESCRIPTION:
"Ancillary-Correlative" study type

PRIMARY OBJECTIVES:

I. To determine whether endogenous metabolomics compounds obtained before cyclophosphamide administration can predict the ratio of 4hydroxycyclophosphamide to cyclophosphamide area under the curve (4HCY/CY AUC).

II. To evaluate mathematic models of CY and mycophenolic acid (MPA) pharmacokinetics and develop mathematic models including these pharmacokinetics, -omics data and clinical outcomes.

SECONDARY OBJECTIVES:

I. To assess if recipients' metabolomics and pharmacokinetics (e.g., CY and its metabolites AUCs) are associated with acute graft versus host disease (GVHD) and other clinical outcomes.

II. To assess the association of the intestinal microbiome with the plasma metabolome, acute GVHD and other clinical outcomes.

III. To obtain donor blood samples at one time pre-transplant and assess if donors' metabolomics are associated with acute GVHD and other clinical outcomes.

EXPLORATORY OBJECTIVE:

I. Donor and recipient germline deoxyribonucleic acid (DNA) isolation and genomic analysis.

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I (PATIENTS RECEIVING A HAPLOIDENTICAL TRANSPLANT): Patients undergo collection of blood prior to transplant, on day 0, days 3-7, day 14, and day 21. Patients also undergo collection of saliva prior to transplant and collection of stool prior to and post-transplant. Donors undergo collection of blood and saliva within 8 weeks prior to donation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo allogeneic hematopoietic cell transplant (HCT) with a haploidentical donor.
* Allogeneic HCT scheduled to treat any underlying disease. Patients with nonmalignant diseases or cancer are eligible
* Scheduled to receive post-transplant cyclophosphamide (any dose, any number of doses, any dosing frequency) as part of their post-graft immunosuppression or GVHD prophylaxis. Patients enrolled on treatment protocols that include post transplant cyclophosphamide (PTCy) but do not include mycophenolate mofetil (MMF) or tacrolimus can participate
* Willingness to:

  * Provide blood
  * Permit medical record review

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the City of Hope Comprehensive Cancer Center and donors.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2027-04-24 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Mathematical models of cyclophosphamide (CY) and mycophenolic acid pharmacokinetics (PK) with t cell effects. | Up to day 21
  Will determine whether readily available patient characteristics influence CY PK using population (pop)PK modeling. Will validate our existing popPK model of CY, 4HCY, and carboxyethylphosphoramide mustard.

SECONDARY OUTCOMES:
Acute GVHD | Up to 4 years
  Cumulative incidence estimates will be calculated with appropriate accounting for competing risks. Adjusted hazard ratios will be estimated via Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine S McCune, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States